CLINICAL TRIAL: NCT00453336
Title: A Phase II Clinical Trial on the Efficacy of Photodynamic Therapy With Porfimer Sodium (Photofrin®) for Malignant and Pre-Malignant Lesions and Condemned Mucosa Syndrome in the Upper Aerodigestive Tract
Brief Title: Photodynamic Therapy With Porfimer Sodium in Treating Patients With Precancerous Lesions, Cancer, or Other Disease of the Aerodigestive Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020618; SCCC-2002103 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20050715 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer; Precancerous/Nonmalignant Condition
Keywords: recurrent squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; oral leukoplakia
MeSH Terms: conditions — Head and Neck Neoplasms; Precancerous Conditions; Squamous Cell Carcinoma of Head and Neck; Leukoplakia, Oral | interventions — Dihematoporphyrin Ether; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Porfimer Sodium; Procedure: Photodynamic Therapy

INTERVENTIONS:
Drug: Porfimer Sodium — Day 1 of Therapy. An IV access (of 20 gauge or larger) is started and 2 mg/kg of Porfimer Sodium (Photofrin®) is given intravenously. Once completed the patient puts on the light protective gear and is sent home.
  Other Names: Photofrin
Procedure: Photodynamic Therapy — Laser Activation. The time of exposure and the power of the laser are computed based on the dosimetry in appendix A using a computed energy dose of 75 to 150 joules, depending on the depth of penetration desired.
  Other Names: Microlens Diffuser P/N 5416

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, precancerous cells and cancer cells are killed.

PURPOSE: This phase II trial is studying the side effects and how well photodynamic therapy with porfimer sodium works in treating patients with precancerous lesions, cancer, or other disease of the aerodigestive tract.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of photodynamic therapy with porfimer sodium in patients with pre-malignant lesions, carcinoma in situ, select superficial squamous cell carcinoma of the oral cavity, oropharynx, or larynx, or condemned mucosa syndrome in the upper aerodigestive tract.
* Determine the safety of this regimen in these patients.

OUTLINE: Patients are stratified according to disease condition (benign vs malignant).

Patients receive porfimer sodium IV over 3-5 minutes on day 1 and laser light activation on day 3 or 4.

After completion of study treatment, patients are followed at 3 and 4 months and then periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Any of the following benign lesions:

    * Localized severe dysplasia, leukoplakia, erythroplakia, or other superficial lesions considered to be pre-malignant
    * Carcinoma in situ
  * Superficial (< 1 cm depth of invasion) squamous cell carcinoma (SCC) of the oral cavity, oropharynx, or larynx

    * T1-T3 disease
    * Meets one of the following criteria:

      * Failed radiation therapy and refused standard salvage surgery
      * Refused radiation therapy and/or surgery as primary therapy
      * No good surgical alternative with acceptable morbidity
  * Condemned mucosa syndrome

    * At least one upper aerodigestive tract pre-malignant lesion, carcinoma in situ, or squamous cell carcinoma previously treated with surgery and/or radiation therapy with the development of another lesion not at the site of the previously treated areas

PATIENT CHARACTERISTICS:

* Creatinine ≤ 2 mg/dL
* AST and ALT ≤ 30% elevated
* Alkaline phosphatase ≤ 30% elevated
* Bilirubin ≤ 1.0 mg/dL
* No contraindication to anesthesia or analgesia
* No porphyria
* No hypersensitivity to porphyrins
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-06; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Civantos, Jr., MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Result] Civantos F. Photodynamic therapy for head and neck lesions in the subtropics. J Natl Compr Canc Netw. 2012 Oct 1;10 Suppl 2:S65-8. doi: 10.6004/jnccn.2012.0179. PMID 23055220

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Photodynamic Therapy : Laser Activation. The time of exposure and the power of the laser are computed based on the dosimetry in appendix A using a computed energy dose of 75 to 150 joules, depending on the depth of penetration desired.
  Porfimer Sodium : Day 1 of Therapy. An IV access (of 20 gauge or larger) is started and 2 mg/kg of Porfimer Sodium (Photofrin®) is given intravenously. Once completed the patient puts on the light protective gear and is sent home.
Period: Overall Study
Arm/Group | Single Arm
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 34
Age, Continuous [Median (Full Range); unit: years] | 66 [30 to 92]
Gender [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 45
Types of Lesions [Number; unit: participants] — The types of lesions participants had at time of enrollment
  participants
    Oral Cavity Lesions | 24
    Layngeal Lesions | 18
    Other Lesions | 3
Pathology [Number; unit: participants]
  Squamous Cell Carcinoma | 22
  Severe Dysplasia | 13
  Carcinoma in situ | 9
  Verrucous Carcinoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Complete or Partial Response 4 Months After Completion of Study Treatment
Description: Number of subjects achieving complete response or partial response to study treatment according to RECIST Criteria version 1.0.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 45
participants | 32

2. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants enrolled experiencing serious adverse events and/or other non-serious events
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 45
participants | 36

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 24/45
Other Adverse Events (participants affected / at risk) | 12/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=45)
Unfortunate Airway Disaster (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Significant Postoperative Pain for Oral Lesions (General disorders) | 23 (23)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=45)
Mild Skin Irritation (Skin and subcutaneous tissue disorders) | 8 (8)
Transient second-degree burn on the back of the hand (Injury, poisoning and procedural complications) | 1 (1)
Inflammatory Reaction from Extravasation of Porfimer Sodium at the Intravenous Site (Injury, poisoning and procedural complications) | 1 (1)
Transient Aspiration (Surgical and medical procedures) | 1 (1)
Temporary edema requiring tracheotomy (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes